CLINICAL TRIAL: NCT06802328
Title: An Intermediate-Size Patient Population Expanded Access Treatment Protocol Evaluating the Safety, Tolerability and Immune Effects of the Nasal Anti-CD3 Monoclonal Antibody Foralumab in Non-Active Secondary Progressive MS Patients Foralumab Nasal
Brief Title: Intermediate-Size Patient Population Expanded Access: Foralumab in Non-Active Secondary Progressive MS Patients
Status: Available | Type: Expanded Access
Sponsor: Tiziana Life Sciences LTD (Industry)
Responsible Party: Sponsor
Other Study IDs: 161148
Record Dates: First submitted 2025-01-23; First posted 2025-01-31 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-03

CONDITIONS: Non-Active Secondary Progressive Multiple Sclerosis
Keywords: multiple sclerosis; non-active secondary progressive multiple sclerosis; MS; expanded access; anti-cd3 monoclonal antibody; foralumab; nasal
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Foralumab TZLS-401 50 µg — Foralumab 50 µg/dosing day for patients who have failed current therapies. Patients will be dosed in 3-week cycles, with foralumab dosing on Days 1, 3 and 5 of the first and second weeks, followed by a "rest week". Patients will receive Day 1 doses of nasal foralumab under supervision at the Center for Clinical Investigation at BWH.

SUMMARY:
This is an open-label, intermediate-size patient population expanded access treatment study utilizing 1 dose level of nasal Foralumab (50 µg/dosing day) with the possibility of increasing to 100 µg/dosing day. The goal of this expanded access clinical trial is to evaluate safety, tolerability, and immune effects of intranasal Foralumab in non-active secondary progressive multiple sclerosis patients. The primary objective is to treat patients who have failed current available therapy. Participants will visit the clinic for testing and follow-up every cycle (3 weeks) while administering the medication at home if able three times weekly.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a common autoimmune disorder affecting young adults, driven by an aberrant T cell response against central nervous system (CNS) antigens. Epidemiologic studies show that approximately 50% of patients are classified as having relapsing-remitting multiple sclerosis (RRMS), while about 35% have SPMS and the remaining 15% have primary progressive MS (PPMS).

Foralumab is a human anti-CD3 monoclonal antibody being developed for the treatment of autoimmune and inflammatory diseases. It is hypothesized that nasal Foralumab will slow disability accumulation and microglial activation measured by PET imaging in non-active SPMS.

Patients will be dosed in 3-week cycles, with Foralumab dosing on Days 1, 3 and 5 of the first and second weeks, followed by a "rest week". This study will assess the safety of nasal Foralumab given over 6 months to non-active secondary progressive MS patients who have failed currently available treatments including the standard of care therapy, Ocrevus (ocrelizumab).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of MS (according to the 2010 McDonald criteria).
* Age 25-75 years old.
* Clinical diagnosis of non-active SPMS, as defined by the absence of relapses for 2 years.
* MRI imaging consistent with a diagnosis of MS at any time point.
* Score on the Expanded Disability Status Scale (EDSS) of 2.5-7.5.
* Have failed standard of care treatment and continued to decline clinically for at least 6 months.
* Adequate hematologic parameters without ongoing transfusion support:

  1. Hemoglobin (Hb) ≥ 9 g/dL
  2. Platelets ≥ 100 x 109 cells/L
* Creatinine ≤ 1.5 x the upper limit of normal (ULN), or calculated creatinine clearance ≥ 60 mL/minute x 1.73 m2 per the Cockcroft-Gault formula.
* Total bilirubin ≤ 2 times the upper limit of normal (ULN) unless due to Gilbert's disease.
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 times ULN.
* QT interval corrected for rate (QTcF) ≤ 470 msec for women and ≤ 450 msec for men on the ECG obtained at Screening
* Negative urine pregnancy test within 7 days prior to the first dose of study therapy for women of child-bearing potential (WCBP), defined as a sexually mature woman who has not undergone a hysterectomy or who has not been naturally postmenopausal for at least 24 consecutive months (i.e., who has had menses any time in the preceding 24 consecutive months). Sexually active WCBP and male patients must agree to use highly effective methods to avoid pregnancy (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) throughout the study and for 90 days after the completion of study treatment.
* Patients whose immunizations are fully up to date at the Screening, according to the assessment of their primary care physician and neurologist.
* Ability to provide written informed consent.

Exclusion Criteria:

* Need for corticosteroid treatment (oral or intravenous) within the past 30 days or anticipated need within 30 days of foralumab therapy initiation.
* Treatment with Ocrevus® (ocrelizumab), Rituxun® (rituximab), Kesimpta® (ofatumumab), Truxima® (rituximab-abbs) within the past 90 days.
* Treatment with Lemtrada® (alemtuzumab) and Mavenclad® (cladribine) within the past 1 year.
* Treatment with chronic immunosuppressives such as interferon, glatiramer acetate, fingolimod, siponimod, dimethyl fumarate or natalizumab within the past 90 days.
* Inability to tolerate nasally administered medications.
* Nasal corticosteroids, nasal antihistamines, nasal flu dosing within the past 30 days, or anticipated need during the study.
* Chronic rhinitis, deviated septum, nasal polyps, history of sinusitis treated within the past 8 months.
* Active COVID-19 disease.
* COVID-19 vaccine within past 10 days or any other vaccine within past 7 days (at dosing).
* Female patient who is pregnant, lactating, breastfeeding, or planning on becoming pregnant during study.
* Female patients of childbearing age will undergo a pregnancy test and be excluded from the study if positive.
* Active malignancy within 5 years.
* Inflammatory bowel disease, rheumatoid arthritis, systemic lupus erythematosus, asthma, or type 1 diabetes.
* Neutropenia or an absolute neutrophil count of < 1,000 cells/mL or other indicators of severe immunosuppression.
* Patients with a history of gadolinium allergy.
* Screening labs outside of the normal range; EBV IgM positive patients with clinical signs will not receive study drug.
* Serious cardiac condition within the last 6 months, such as uncontrolled arrhythmia, myocardial infarction, unstable angina, or heart disease defined by the New York Heart Association (NYHA) Class III or Class IV or hereditary long QT syndrome.
* Concomitant medication(s) that may cause QTc prolongation or induce Torsades de Pointes, except for antimicrobials that are used as standard of care to prevent or treat infections and other such drugs that are considered by the Investigator to be essential for patient care.
* Patients who test positive for human immunodeficiency virus (HIV), hepatitis B virus surface antigen (HBsAg), or hepatitis C virus (HCV) at the Screening Visit.
* A recent clinically significant active infection requiring treatment with antibiotics or other anti-infective agents within the past 15 days.
* Patients whose immunizations are not fully up to date at the Screening Visit, as assessed by their primary care physician and neurologist.
* Any other medical intervention or other condition which, in the opinion of the Principal Investigator, could compromise adherence to study requirements or confound the interpretation of study results.
* Unable or unwilling to comply with protocol requirements.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States